CLINICAL TRIAL: NCT03986905
Title: A Randomized, Double Blind, Placebo-Controlled Phase 3 Study of the Safety and Efficacy of DPI-386 Nasal Gel on Ocean Going Vessels for the Prevention and Treatment of Nausea Associated With Motion Sickness
Brief Title: The Prevention and Treatment of Nausea Associated With Motion Sickness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DPI-386-MS-21
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A double-dummy design will be used to mask the treatment assignment. A double-dummy design will be used to mask the treatment assignment. A designated independent (unblinded) applicator will administer all patch application and removal, including an opaque waterproof bandage cover over the patch, to further prevent unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Scopolamine Nasal Gel (Experimental): DPI-386 Nasal Gel + placebo patch
  Interventions: Drug: Scopolamine Nasal Gel; Other: Placebo
- Placebo (Placebo Comparator): placebo nasal gel + placebo patch
  Interventions: Other: Placebo
- TDS Patch (Active Comparator): placebo nasal gel + TDS patch
  Interventions: Drug: Scopolamine Nasal Gel; Other: Placebo

INTERVENTIONS:
Drug: Scopolamine Nasal Gel — All subjects will receive both a patch and nasal gel: DPI-386 Nasal Gel + placebo patch, placebo nasal gel + placebo patch, or placebo nasal gel + TDS patch.
  Other Names: Scopolamine Patch
  Arms: Scopolamine Nasal Gel; TDS Patch
Other: Placebo — placebo nasal gel + placebo patch
  Other Names: Placebo Patch and Placebo Nasal Gel

SUMMARY:
This single-site Phase 3 clinical trial is a randomized, double-blind, placebo-controlled study to identify the safety and efficacy of a repeated-dose regimen of DPI 386 nasal gel (intranasal scopolamine gel) for the prevention and treatment of nausea associated with motion sickness. The study will be conducted aboard an ocean going vessel to obtain data in a real world environment. The study will have three arms: DPI-386 nasal gel, placebo nasal gel, and TDS patch (1.5 mg/72 hours), the current standard of care for the treatment of motion sickness. The study will include 100 subjects per arm, for a total of 300 subjects (n=300). Multiple voyages with the same vessel will be used until the required enrollment is completed. A double dummy design will be used to mask the treatment assignment. All subjects will receive both a patch and nasal gel randomized to one of the following three arms: DPI-386 Nasal Gel + placebo patch, placebo nasal gel + placebo patch, and placebo nasal gel + TDS patch.

DETAILED DESCRIPTION:
The investigational product will be administered using a delivery device comprised of: (a) a vial prefilled with DPI-386 Nasal Gel or placebo nasal gel, and (b) a nasal gel pump attached to the vial during the manufacturing process. Each 0.12 gram of the gel contains 0.2 mg of scopolamine HBr as the active ingredient along with the excipients sodium citrate, citric acid, sodium metabisulfite, glycerin, benzalkonium chloride, polyvinyl alcohol and purified water. The DPI 386 Nasal Gel is formulated to contain 0.2 mg scopolamine HBr per 0.12 g dose, with each dose therefore described as "0.2 mg / 0.12 g". The placebo nasal gel product is the same but does not contain scopolamine HBr. Each vial of DPI 386 Nasal Gel or placebo nasal gel is a multi-dose product, sufficient for three days of dosing (two doses per day). Each pumping action is designed to deliver a single 0.12 g dose. Each vial/delivery device must be primed by the subject prior to first dose delivery for that vial. Each time a new bottle is used, it needs to be initially primed with 5 actuations. The 6th actuation is the first dose and subsequent actuations are doses 2-6 of that bottle. No re-priming is needed at all. Subjects will be trained in priming by research staff, and all priming will be performed under supervision by the research staff. All subjects will self-administer the nasal gel twice daily over the three day treatment period, with no more than two doses every 24 hours, unless a third dose is deemed necessary by the PI or qualified designee, and the two daily doses separated by a minimum of six hours ± 15 minutes

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated Informed Consent Form (ICF).
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18 to 59 (inclusive).
* At least minimally susceptible to provocative motion as evidenced by a minimum score of 3.0 on the Motion Sickness Susceptibility Questionnaire (MSSQ).
* In good general health as evidenced by medical history with no recent history or current diagnosis of uncontrolled clinical problems as assessed by the Principal Investigator (PI) or qualified designee.
* Ability to take intranasal medication and willingness to adhere to the study schedule and time constraints.
* For females of child-bearing potential: willingness to provide a urine sample for the hCG pregnancy test. The test must be negative within seven days of Treatment Day 1.
* Agreement to adhere to the following lifestyle compliance considerations:
* Refrain from consumption of grapefruit and any substance containing grapefruit for seven days prior to, during, and for seven days after the three Treatment Days.
* Abstain from alcohol for 24 hours prior to first dose of study medication and during the three Treatment Days.

Exclusion Criteria:

* Pregnancy, lactation, or positive urine pregnancy test within seven days of Treatment Day 1.
* Known allergic reactions to scopolamine or other anticholinergics.
* Currently prescribed any of the following medication types and used within the specified washout periods below:
* any form of scopolamine (including Transderm Scop®) (washout 5 days)
* belladonna alkaloids (washout 2 weeks),
* antihistamines (including meclizine) (washout 2 weeks),
* tricyclic antidepressants (washout 2 weeks),
* muscle relaxants (washout 4 days) and
* nasal decongestants (washout 4 days)
* Hospitalization or significant surgery requiring hospital admittance within the past six months.
* Treatment with another investigational drug or other intervention within the past 30 days.
* Having donated blood or plasma or suffered significant blood loss within the past 30 days.
* Having any of the following medical conditions within the last two years or if any of the following medical conditions were experienced more than two years ago and are deemed clinically significant by the PI or qualified designee:

  1. Significant gastrointestinal disorder, asthma, or seizure disorders.
  2. History of vestibular disorders.
  3. History of narrow-angle glaucoma.
  4. History of urinary retention problems.
  5. History of alcohol or drug abuse.
  6. Nasal, nasal sinus, or nasal mucosa surgery.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
The efficacy endpoint is incidence of subjects who developed motion sickness and request further treatment during an 8 hour voyage | During three consecutive days
  The efficacy endpoint is incidence of subjects who developed motion sickness and request further treatment with Rescue medication during an 8 hour voyage on Treatment Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Helton, Study Director — Repurposed Therapeutics, Inc.
Locations (1):
- Collaborative Neuroscience Network, LLC, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
In publication and CSR.